CLINICAL TRIAL: NCT05163561
Title: A Phase III, Double Blind, Randomized, Active Controlled Study to Evaluate Safety and Immunogenicity of Inactivated Adjuvanted Polio Vaccine in Comparison With Licensed Inactivated Poliovirus Vaccine
Brief Title: Evaluation of Safety and Immunogenicity of Inactivated Adjuvanted Polio Vaccine in Comparison With Licensed Inactivated Poliovirus Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Serum Institute of India Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IPV:02
Record Dates: First submitted 2021-12-03; First posted 2021-12-20 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Intervention Model Description: Study participants aged 6 to 8 weeks will be enrolled and randomized into 1:1:1:1 ratio to receive either the SII inactivated Salk polio vaccine (adsorbed) from one of the three lots (Lot A or Lot B or Lot C) or the Sii licensed inactivated poliovirus vaccine (IPV).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is designed as a double-blind (observer blind) study. Observer-blind means that during study, the participants and the study personnel responsible for the evaluation of any study endpoints (e.g. safety and immunogenicity) will be unaware of the IP administered. The IP preparation and administration will be done by designated unblinded personnel who will not participate in any of the clinical study evaluations. Unblinded study personnel will prepare/reconstitute the IP out of view of the participant as well as the site staff. Considering the fact that the IP are likely to have distinct appearances, even when drawn into syringes, the syringes will be masked with an opaque wrapping before administration. After administration, the unblinded study personnel will complete accountability label on the carton and store the used products at designated area.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SII Inactivated Salk Polio Vaccine (Adsorbed) Lot A (Experimental): SII Inactivated Salk Polio Vaccine (Adsorbed) Lot A
  Interventions: Biological: SII Inactivated Salk Polio Vaccine (Adsorbed) - Lot A
- SII Inactivated Salk Polio Vaccine (Adsorbed) Lot B (Experimental): SII Inactivated Salk Polio Vaccine (Adsorbed) Lot B
  Interventions: Biological: SII Inactivated Salk Polio Vaccine (Adsorbed) - Lot B
- SII Inactivated Salk Polio Vaccine (Adsorbed) Lot C (Experimental): SII Inactivated Salk Polio Vaccine (Adsorbed) Lot C
  Interventions: Biological: SII Inactivated Salk Polio Vaccine (Adsorbed) - Lot C
- Sii Licensed IPV (Active Comparator): Sii Licensed IPV
  Interventions: Biological: Sii Licensed IPV

INTERVENTIONS:
Biological: SII Inactivated Salk Polio Vaccine (Adsorbed) - Lot A — SII Inactivated Salk Polio Vaccine (Adsorbed) produced by Serum Institute of India Pvt. Ltd., is a sterile suspension of three types of inactivated poliovirus: Type 1 (Mahoney), Type 2 (MEF-1), and Type 3 (Saukett). It is a highly purified, adjuvanted reduced antigen content of inactivated poliovirus vaccine.
  Arms: SII Inactivated Salk Polio Vaccine (Adsorbed) Lot A
Biological: SII Inactivated Salk Polio Vaccine (Adsorbed) - Lot B — SII Inactivated Salk Polio Vaccine (Adsorbed) produced by Serum Institute of India Pvt. Ltd., is a sterile suspension of three types of inactivated poliovirus: Type 1 (Mahoney), Type 2 (MEF-1), and Type 3 (Saukett). It is a highly purified, adjuvanted reduced antigen content of inactivated poliovirus vaccine.
  Arms: SII Inactivated Salk Polio Vaccine (Adsorbed) Lot B
Biological: SII Inactivated Salk Polio Vaccine (Adsorbed) - Lot C — SII Inactivated Salk Polio Vaccine (Adsorbed) produced by Serum Institute of India Pvt. Ltd., is a sterile suspension of three types of inactivated poliovirus: Type 1 (Mahoney), Type 2 (MEF-1), and Type 3 (Saukett). It is a highly purified, adjuvanted reduced antigen content of inactivated poliovirus vaccine.
  Arms: SII Inactivated Salk Polio Vaccine (Adsorbed) Lot C
Biological: Sii Licensed IPV — Poliomyelitis Vaccine (Inactivated), produced by Serum Institute of India Pvt. Ltd., is a sterile suspension of three types of inactivated poliovirus: Type 1 (Mahoney), Type 2 (MEF-1), and Type 3 (Saukett). Poliomyelitis Vaccine (Inactivated) is a highly purified, inactivated poliovirus vaccine.
  Arms: Sii Licensed IPV

SUMMARY:
This Phase III study has been designed to compare the SII Inactivated Salk Polio Vaccine (Adsorbed) with Sii licensed IPV by testing the vaccine in infants (three doses administered 4 weeks apart, starting at 6-8 weeks of age) in order to demonstrate the non-inferiority in the induction of specific poliovirus neutralizing antibody (PVNA) to poliovirus type 1, type 2 and type 3 by these vaccines. The study will also evaluate lot-to-lot consistency in the manufacture of SII Inactivated Salk Polio Vaccine (Adsorbed) by demonstrating equivalence in the induction of PVNA across three production lots.

DETAILED DESCRIPTION:
The study is designed as a double-blind, randomized, active-controlled Phase III study with four groups of infants (n=268 per group) receiving either SII Inactivated Salk Polio Vaccine (Adsorbed) from the three lots or Sii licensed IPV.

Participants will be screened for eligibility with their parental consent and will be selected for the study according to inclusion and exclusion criteria. A total of 1072 participants will be enrolled.

Following vaccination, enrolled participants will remain in the clinic for at least 30 minutes for observation. During this time, they will be closely monitored for any immediate adverse events. Safety will be evaluated by active surveillance for solicited adverse events over the 4-day period after each vaccination in all participants. In addition, surveillance for unsolicited AEs and SAEs will be carried out over the period from first vaccination and 28 days after the third vaccination in all participants.

The immunogenicity will be assessed by measuring the PVNA to poliovirus type 1, type 2 and type 3 using a standardized microneutralization test in the sera samples of the participants.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants as established by medical history and clinical examination before entering the study
2. Age: 6-8 weeks at the time of enrolment
3. Parental ability and willingness to provide informed consent
4. Parent who intends to reside in the area with the infant during the study period

Exclusion Criteria:

1. Presence of fever on the day of enrolment [Temporary exclusion criteria].
2. Acute disease at the time of enrolment [Temporary exclusion criteria].
3. Prior receipt or intent to receive OPV/IPV/IPV containing vaccines during the study period.
4. OPV vaccination or known exposure to poliovirus (wild or vaccine derived) in household (living together) within 3-months prior to inclusion or planned during the study.
5. Presence of significant malnutrition (weight-for-height z-score < -3SD median)
6. Known or suspected impairment of immunological function based on medical history and physical examination.
7. Presence of any systemic disorder (cardiovascular, pulmonary, hepatic, renal, gastrointestinal, hematological, endocrine, immunological, dermatological, neurological, cancer, or autoimmune disease) as determined by medical history and / or physical examination which would compromise the participant's health or is likely to result in nonconformance to the protocol.
8. A known sensitivity or allergy to any components of the Investigational Product.
9. Receipt of immunoglobulin therapy and / or blood products since birth or planned administration during the study period
10. Planned concurrent participation in another clinical study at any point throughout the entire study period

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1072 (Actual)
Dates: Start 2022-01-09 (Actual); Primary Completion 2023-04-29 (Actual); Study Completion 2023-04-29 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with type-specific seroconversion | Day 28 after third vaccination
  Percentage of participants with type-specific seroconversion* on Day 28 after the third vaccination for SII Inactivated Salk Polio Vaccine (Adsorbed) and Sii Licensed IPV

SECONDARY OUTCOMES:
Geometric Mean Titers | Day 28 after third vaccination
  Type-specific geometric mean titers on day 28 after the third vaccination of three cGMP lots of SII Inactivated Salk Polio Vaccine (Adsorbed) and Sii Licensed IPV.
Reverse cumulative distribution curves of antibody titers | pre-vaccination and 28 days after third vaccination
  Type-specific reverse cumulative distribution curves of antibody titers on pre-vaccination and 28 days after third vaccination of three cGMP lots of SII Inactivated Salk Polio Vaccine (Adsorbed) and Sii Licensed IPV.
Percentage of participants with type-specific seroprotection | Day 28 after the third vaccination
  Percentage of participants with type-specific seroprotection (titers ≥ 8) on Day 28 after the third vaccination of three cGMP lots of SII Inactivated Salk Polio Vaccine (Adsorbed) and Sii Licensed IPV.
Percentage of participants with type-specific post-vaccination titers ≥ 4-fold above the estimated titer of maternal antibody | Day 28 after the third vaccination
  Percentage of participants with type-specific post-vaccination titers ≥ 4-fold above the estimated titer of maternal antibody on day 28 after the third vaccination of three cGMP lots of SII Inactivated Salk Polio Vaccine (Adsorbed) and Sii Licensed IPV.

CONTACTS AND LOCATIONS:
Overall Officials: K Zaman, MD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh (ICDDR,B), Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kulkarni PS, Zaman K, Desai SA, Bharati S, Goswami DR, Sharmeen AT, Rana S, Haque W, Khandelwal A, Manney S, Tyagi P, Gairola S, Zade JK, Pisal SS, Dhere RM, Poonawalla CS, Lamberigts C, Parulekar V, Potey AV. Safety and immunogenicity of a reduced-dose inactivated poliovirus vaccine versus a full-dose inactivated poliovirus vaccine in infants in Bangladesh: a double-blind, non-inferiority, randomised, controlled, phase 3 trial. Lancet Infect Dis. 2025 Oct;25(10):1128-1137. doi: 10.1016/S1473-3099(25)00215-4. Epub 2025 Jun 9. PMID 40505670